CLINICAL TRIAL: NCT04468386
Title: Specimen Collection Study Protocol; Internal Biomerica Normal Specimen Collection and Banking for Use in COVID-19 Serological Product Development
Brief Title: Specimen Collection Study Protocol
Status: Completed | Type: Observational
Sponsor: Biomerica (Industry)
Responsible Party: Sponsor
Other Study IDs: CV19-Col-004
Record Dates: First submitted 2020-07-08; First posted 2020-07-13 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2020-07

CONDITIONS: Focus in on Collecting Paired Specimens for Matrix Equivalency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, Plasma and Dried Blood Spots (DBS - whole blood dried on filter paper). Serum and Plasma will be retained the DBS will be depleted and not retained
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The specimens collected will be used to evaluate matrix equivalency in an immunoassay in development for the detection of IgG or IgA or IgM antibodies to SARS - CoV2 in human serum. These reagents are for in vitro diagnostic use only.

DETAILED DESCRIPTION:
The objective of this study is to acquire paired serum, plasma and whole blood collected on a collection card from subjects with no known history of COVID-19 infection. The specimens will be collected at Biomerica in Irvine CA for specimen collection, banking, and matrix equivalency studies for projects in development at Biomerica for detection to IgG or IgA or IgM antibodies to Sars-CoV2 antibodies. Subject will also be asked to self-collect a nasal swab for COVID-19 PCR

ELIGIBILITY:
Inclusion Criteria:

* Aged 21 and older
* Able to read, speak, and understand English
* Must weigh a minimum of 110 pounds
* Willing and able to donate 20 mLs of whole blood via venipuncture. [approximately ˂ 2 tablespoons]
* Willing and able to donate 0.040 mLs of whole blood via fingerstick
* Willing and able to sign the informed consent (self or authorized representative)
* Willing and able to self-collect a nasal swab per the provided instruction shee

Exclusion Criteria:

* Aged less than 21 years old
* Unable to provide consent.
* Unable to donate blood via venipuncture and fingerstick.
* Unable to self-collect a nasal swab

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of subjects identified as meeting the inclusion/exclusion criteria from Biomerica employees and/or friends and family of Biomerica's employees. There will be no outside advertising or recruiting. All subjects must be willing to sign the informed consent and undergo the venipuncture and finger stick blood collection process and perform the nasal swab collection.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Matrix Equivalency | 1 day
  This study is designed to collect specimens to support specimen matrix equivalency in an in vitro diagnostic assay for the detection of COVID-19 antibodies.
  Additionally, specimens collected via finger stick will be used to validate a whole blood collection card that could be used in the field by trained professionals and sent back to central reference laboratories for testing.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Laderman, Ph.D., Principal Investigator — Biomerica, Inc.
Locations (1):
- Biomerica, Inc., Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No